CLINICAL TRIAL: NCT01738061
Title: A Multidimensional Lifestyle Intervention to Reduce the Risk of Metabolic Disorders in Older Workers in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government)
Responsible Party: Principal Investigator, Alan C. Tsai, Ph. D., professor, Asia University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MM-WHP-99
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Metabolic Disorder
Keywords: Older workers; Multidimensional intervention; Worksite health promotion; Taiwan
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reference group (No Intervention): They continued their daily routine.
- Multidimensional lifestyle intervention (Experimental): The multidimensional lifestyle intervention program received motivational activities to improve awareness of the impact of lifestyle on chronic diseases and the importance of self-health management.
  Interventions: Behavioral: Multidimensional lifestyle intervention

INTERVENTIONS:
Behavioral: Multidimensional lifestyle intervention — Lecture series to increase awareness of the relationship of lifestyle to chronic diseases Individualized review and discussion to understand own health problems Biweekly group meetings to stimulate motivation and exchange ideas
  Arms: Multidimensional lifestyle intervention

SUMMARY:
The study was aimed to evaluate the effectiveness of a multidimensional worksite intervention program to reduce the severity of metabolic disorders in older workers in Taiwan.

DETAILED DESCRIPTION:
The investigators conducted a quasi-experiment in older workers from three worksites in southern Taiwan.

* Qualified subjects were assigned to the intervention or the reference group according to their availability to take part in study activities.
* A researcher reviewed the health record and discussed with the subject about his/her health status.
* Subjects in the intervention group received lifestyle interventions. The activities included motivational presentations to increase awareness of own health problems and the role of lifestyle in the etiology of non-communicable chronic diseases.
* Subjects were organized into small groups to have biweekly meetings to share experiences, stimulate mutual encouragement and to overcome obstacles.
* Anthropometric and biochemical indicators were measured at baseline and endpoint (week 24).

ELIGIBILITY:
Inclusion Criteria:

* full-time worker
* aged 50 years or older
* willing to complete a screening questionnaire
* sign a study consent

Exclusion Criteria:

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-01; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in anthropometric and srum biochemical indicators. | At baseline (week 0) and endpoint (week 24) of the intervention
  Body weight (BW), body height, waist circumference, Body mass index (BMI), arterial blood pressure (BP), serum total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG) and glycosylated hemoglobin (HbA1c) concentrations

SECONDARY OUTCOMES:
Lifestyle factors | At baseline (week 0) and endpoint (week 24) of the intervention
  Physical activity, food consumption frequency and self-reported sleep and sedentary hours.

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Tsai, PhD, Principal Investigator — Department of Healthcare Administration, Asia University